CLINICAL TRIAL: NCT05211167
Title: A Multicenter, Randomized, Parallel-controlled Phase III Trial Comparing the Efficacy and Safety of Recombinant Erythropoiesis Stimulating Protein Injection (CHO Cell) With Ipbio in Maintenance Therapy in Hemodialysis Patients With Anemia in Chronic Renal Failure
Brief Title: Phase III Clinical Study of Recombinant Erythropoiesis Stimulating Protein Injection (rESP) in the Treatment of Anemia in Hemodialysis Patients With Chronic Renal Failure
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSS-SSS06-HD-III-01
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Kidney Failure, Chronic; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Intravenous administration, maintaining the same dose and frequency administrated in the sceening period, for 32 weeks
  Interventions: Drug: Human Erythropoiesis Injection (CHO cell)
- Group B (Experimental): Intravenous administration,50μg, once every two weeks, for 32 weeks
  Interventions: Drug: Recombinant Erythropoiesis Stimulating Protein Injection(CHO cell)

INTERVENTIONS:
Drug: Human Erythropoiesis Injection (CHO cell) — Human Erythropoiesis Injection (CHO cell) is a recombinant human erythropoietin with the same biological effects as natural erythropoietin
  Arms: Group A
Drug: Recombinant Erythropoiesis Stimulating Protein Injection(CHO cell) — rESP is a high glucose medium and long-acting recombinant protein products, containing 165 amino acids by adding 3 glycosylation sites
  Other Names: rESP
  Arms: Group B

SUMMARY:
To verify the efficacy of recombinant erythropoiesis stimulating protein injection (CHO cell) in hemodialysis patients with chronic renal failure anemia maintenance treatment is not inferior to yibio.

DETAILED DESCRIPTION:
In this phase 3, open label, active comparator parallel controlled study, patients were randomly assigned to two study groups: one active comparator control group (Human Erythropoietin Injection , maintaining the same dose and frequency administrated in the sceening period ), and experimental groups (50μg, once every two weeks). All the patients were administered intravenously for 32 weeks and were evaluated the efficacy, safety and pharmacokinetic characteristics. During the whole study period, dosage adjustment was not allowed in the first 4 weeks, while in the remaining trial period dosage adjustment was allowed once every two weeks if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer as a subject must understand the study procedure and sign the informed consent form;
* 18 years old ≤ age ≤ 75 years old when sign ICF, gender is not limited;
* Patients diagnosed with chronic renal failure anemia were receiving maintenance hemodialysis for at least 3 months and 2-3 times a week; The dialysis frequency was stable and there was no change in the dialysis plan throughout the study period;
* Before enrollment, patient being treated short-acting EPO stabilization therapy for at least 12 weeks, the average concentration of hemoglobin in the screening period is in the range of 100~120 g/L (including both ends), and the difference is less than 10g/L;
* Iron status and dialysis status were evaluated within 4 weeks before enrollment to meet the following requirements:

Transferrin saturation (TSAT) ≥20% and serum ferritin (SF) ≥200 μg/L; Dialysis parameters: urea clearance index spKt/V≥1.2;

* Subjects agree to use reliable contraceptives by themselves and their spouses from the screening period to within 3 months after the end of the study;

Exclusion Criteria:

* Allergic to the investigational drug or any ingredient in the investigational drug or has had a severe allergic reaction to the drug in the past;
* Except of renal anemia, there are other diseases that cause chronic anemia (such as sickle cell anemia, myelodysplastic syndrome, hematological malignancies, myeloma, hemolytic anemia, pure red blood cell aplastic anemia), blood systemic disease or coagulopathy;
* Patients who have received or plan to have a kidney transplant during the study period, or who plan to have other surgical procedures during the study period (mainly major surgeries, except those with low blood loss that do not affect Hb concentration);
* Patients with acute or chronic blood loss (such as upper gastrointestinal bleeding, etc.) within 3 months prior to enrollment were excluded from the scope of hemorrhage caused by minor surgeries such as temporary vascular access required by clinical medical procedures;
* Patiernts who was suffering from malignant hypertension or poor control of blood pressure (systolic blood pressure >180 mmHg or diastolic blood pressure >100 mmHg);
* The following conditions (including but not limited to) occurred in the laboratory examination during the screening period, and the investigator judged that the participants were not eligible for inclusion: a) Patients who were positive for HBsAg, anti-HIV, anti-HCV, and Treponema pallidum antibodies; b) The aspartate aminotransferase or alanine aminotransferase is greater than 3 times the upper limit of normal; c) Serum albumin < 35g/L;
* Patiernts who was suffering from severe secondary hyperparathyroidism (sustained blood iPTH/PTH >1000 ng/L);
* Patients with previous thromboembolic disease (excluding luminal infarction), history of severe hematopoietic system, and high clotting tendency;
* Patiernts with severe cardiovascular and cerebrovascular disease, severe or unstable coronary artery disease, heart failure (NYHA class III or IV), temporary vascular access, or myocardial infarction or stroke within 3 months before enrollment;
* A history of malignant neoplasms, except for: basal cell or squamous cell carcinoma of the skin determined to be cured or no recurrence within 5 years, with radical excision, or carcinoma in situ at any site;
* The researchers identified those with severe infectious disease or chronic, uncontrolled inflammation within the first four weeks of enrollment;
* All epilepsy or epilepsy history except of childhood febrile seizures, post-traumatic or abstinence single seizures;
* Those who have received androgen therapy or who have received blood transfusion therapy within the past 8 weeks before enrollment;
* Patients who had a pacemaker for more than 5 years; If no more than 5 years of cardiac pacemaker working status assessment and test unqualified;
* 3 months as a subject to participate in other new drug clinical trials or to the group when the withdrawal time is shorter than the five half-life of the test drug (whichever is the longest of the two);
* Subjects were in the middle of pregnancy or lactation at the time of enrollment;
* Alcohol, drug or drug addicts;
* Other conditions that may not be suitable for the study as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
hemoglobin concentration | 25th-32nd week
  the amount of change in mean Hb concentration compared with baseline Hb concentration during the evaluation period

SECONDARY OUTCOMES:
maintenance rate | 25th-32nd week
  the proportion of subjects whose average Hb concentration remained within the target range during the evaluation period
proportion of subjects | for 32 weeks
  the proportion of subjects whose range of dose adjustments decreased or increased by 25% still did not reach 100-120 g/L (both ends)
proportion of times | 25th-32nd week
  the proportion of times the measured Hb concentration remains within the target range during the subject evaluation period
average weekly dose | 25th-32nd week
  the average weekly dose of the drug during the evaluation period
average hemoglobin concentration | 25th-32nd week
  the mean Hb concentration during the evaluation period
mean reticulocyte count | 25th-32nd week
  changes in mean values of reticulocyte compared to baseline values during the evaluation period
mean red blood cell count | 25th-32nd week
  changes in mean values of red blood cell count compared to baseline values during the evaluation period
adverse events | for 32 weeks
  the type, proportion and severity of adverse events
number of dose adjustments | for 32 weeks
  the number of dose adjustments used by the subject during the treatment and evaluation period
the ratio of subjects who are adjusted | for 32 weeks
  the ratio of subjects who are adjusted during the treatment and evaluation period
incidence of Human Erythropoietin antibodies and anti-rESP antibodies | for 32 weeks
  incidence of Human Erythropoietin antibodies and anti-rESP antibodies
Maximum Plasma Concentration (Cmax) | for 32 weeks
  the Cmax of rESP in patients with long-term medication
Area Under the Curve (AUC) | for 32 weeks
  the AUC of rESP in patients with long-term medication

CONTACTS AND LOCATIONS:
Overall Officials: XiangMei Chen, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided